CLINICAL TRIAL: NCT03143647
Title: Influence of Therapeutic Magnesium on Platelet Function Testing
Brief Title: Magnesium and Platelet Function Testing
Acronym: MgCedVD
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Dieter Mesotten, MD, Ziekenhuis Oost-Limburg
Other Study IDs: CTU2017140
Record Dates: First submitted 2017-04-26; First posted 2017-05-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Eclampsia Preeclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: * Female
  * Over 18 years of age
  * American Society of Anesthesiologists physical fitness scale 1
  * Not pregnant
  Interventions: Other: Collect a study-specific blood sample of healthy subjects
- Case: * Female
  * Pregnant with possible pre-eclampsia
  * Over 18 years of age
  * American Society of Anesthesiologists physical fitness scale 1
  Interventions: Other: Collect a study-specific blood sample of healthy subjects

INTERVENTIONS:
Other: Collect a study-specific blood sample of healthy subjects — One heparin tube (4ml) and one hirudin tube (4ml) blood sample will be collected through standard venipuncture. After applying a tourniquet with moderate pressure around the arm of the patient's choice, skin will be disinfected over a suitable vein in the elbow or fore-arm. A hirudin and a heparin tube will be filled with venous blood through a single puncture with a 22 Ga needle (manufacturer, location). After release of the tourniquet, bleeding will be stopped by applying local pressure for 5 minutes with a sterile gauze.
  Other Names: Collect an extra blood sample of pregnant woman during a routine control with an already planned blood sample collection

SUMMARY:
Magnesium has built up the reputation of a 'natural calcium antagonist'. However, the exact effect of magnesium on coagulation and more specifically on platelet function is still disputed. An important discrepancy between in vivo and in vitro studies exists. Magnesium has thus been reported to antagonize platelets in some studies, and to stimulate platelets in other studies. Current evidence seems to point in the direction of a general antagonization of aggregation and coagulation.

Intravenous magnesium is often administered in pre-eclampsia as seizure prophylaxis. Therapeutic regimens usually consist of an intravenously administered loading dose (2-3 grams) and a maintenance infusion, targeting a plasma level of 2-3 mmol/L. Therapeutic drug monitoring is needed, as magnesium toxicity is an important concern.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent
* Over 18 years of age (and younger or equal to 50 years of age) and able to provide legally binding consent
* American Society of Anesthesiologists physical fitness scale 1 (non smoker, no or minimal alcohol use, ..)

Exclusion Criteria:

* Chronic disease
* Chronic medical therapy (other than oral contraception)
* Pregnancy
* ASA 2 or higher
* Known coagulation or aggregation disorders
* Use of COX-inhibitors in the last 10 days
* Contra-indications for venipuncture

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Females over 18 years of age (and younger or equal to 50 years of age) that meet the American Society of Anesthesiologists physical fitness scale 1 (non smoker, no or minimal alcohol use, ..)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
PAC-t-UB test results | 4 months
  The main endpoint of this study is the Platelet Activation Test in Unprocessed Blood (PAC-t-UB).

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Mesotten, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No